CLINICAL TRIAL: NCT02499549
Title: A Randomised, Parallel Group Clinical Trial to Assess the Efficacy, Safety and Acceptability of a Surfactant Based Lotion in the Treatment of Head Louse Infection.
Brief Title: Two Treatment Regimens of Cocamide DEA Lotion for Head Lice
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Medical Entomology Centre (Industry)
Collaborators: Riemann a/s (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTRL02
Record Dates: First submitted 2015-07-10; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Pediculosis; Head Louse Infestation
MeSH Terms: conditions — Lice Infestations | interventions — coconut diethanolamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10% Cocamide diethanolamine 8 hours (Experimental): Cocamide DEA topical lotion applied 8 hours/overnight with drying
  Interventions: Drug: cocamide diethanolamine
- 10% Cocamide diethanolamine 2 hours (Experimental): Cocamide DEA topical lotion applied 2 hours with drying, repeated after 7 days
  Interventions: Drug: cocamide diethanolamine

INTERVENTIONS:
Drug: cocamide diethanolamine — 10% Cocamide DEA aqueous lotion is applied directly to dry hair and is washed off with water only
  Other Names: lauramine diethanolamine

SUMMARY:
To assess the efficacy and safety of 10% Cocamide DEA using two treatment regimens in the eradication of head lice. To assess the ability of each treatment regimen to kill all viable ova and to assess patient acceptability of the product in use

DETAILED DESCRIPTION:
A previous study found that a formulation of 10% cocamide diethanolamine (DEA) aqueous lotion showed some efficacy to eliminate head louse infestation but that the treatment regimen was inadequate to kill all lice or louse eggs. This study has been designed to compare two different application regimens that have been shown effective in vitro.

A planned total of 120 patients who, following examination, are found to suffer from active head lice infestation will be recruited to the trial. The patient will be treated with 10% cocamide DEA lotion using the appropriate treatment regimen according to the randomization code from a pre-prepared listing in balanced blocks of 12.

Group 1: 10% cocamide DEA is applied directly to dry hair, the excess water evaporated off using a hair dryer and is then left for 8 hour/overnight before washing off with clean water.

Group 2: 10% cocamide DEA is applied directly to dry hair, the excess water evaporated off using a hair dryer and is then left for 2 hours before washing off with clean water. A follow up treatment is given after 7 days.

Treatments will be applied by experienced investigators throughout the study. Assessments will be made by other investigators unaware of the treatment regimen used.

After treatment (day 0), follow up assessments will be performed on days 4, 8,11 then again at day 14 after which they will leave the study. Any adverse events or side effects from the treatments will be monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over the age of 4 who are found to have a head louse infection.
* Patients who give written informed consent and, if the patient is under 16 years of age, whose guardian gives written informed consent to participate in the study.
* Available for the duration of study i.e. 15 days.

Exclusion Criteria:

* Patients with a known sensitivity to paraben preservatives.
* Patients who have been treated with other head lice products within the last 2 weeks.
* Patients who have undergone a course of antibiotic treatment within the last 4 weeks.
* Patients who have any persistent skin disorder of the scalp (i.e. eczema, chronic dermatitis, psoriasis).
* Patients whose hair has been bleached, colour treated or permed within the last 4 weeks.
* Patients who have participated in another clinical trial within 1 month prior to entry to this study.
* Patients who have already participated in this clinical trial.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 1999-10; Primary Completion 1999-12 (Actual); Study Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
Successful elimination of infestation | 14 days
  No evidence of active head lice infestation 14 days after enrolment

SECONDARY OUTCOMES:
Number of participants with treatment related adverse events as a measure of safety | 14 days
  No treatment related adverse events following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ian F Burgess, Principal Investigator — Medical Entomology Centre